CLINICAL TRIAL: NCT00788190
Title: Treatment of Distal Radius Fractures in Elderly Patients, a Randomized Controlled Trial
Brief Title: Treatment of Distal Radius Fractures in Elderly Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The inclusion/Exclusion criteria was too strict which restricted recruitment
Sponsor: Hand and Upper Limb Clinic, Canada (Network)
Collaborators: LHRI- Lawson Health Research Institute (Unknown)
Responsible Party: Dr. Joy MacDermid, Associate Professor, St. Joseph's hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LHRI 001
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2008-11

CONDITIONS: Distal Radius Fractures
Keywords: Distal Radius Fracture; Elderly; Prospective randomized trial; Outcomes; Pain and Function; Surgical Vs. conservative management; Fractures with borderline alignment
MeSH Terms: conditions — Wrist Fractures; Pain | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery (Other): Surgical intervention to reduce Distal Radius Fracture
  Interventions: Procedure: Distal Radius Fracture Reduction
- Conservative Treatment (Other): Conservative treatment of Distal Radius Fractures
  Interventions: Other: Conservative Management

INTERVENTIONS:
Procedure: Distal Radius Fracture Reduction — Surgical Intervention to Reduce Distal Radius Fracture
  Other Names: Distal Radius Reduction
  Arms: Surgery
Other: Conservative Management — Conservative management of Distal Radius Fractures
  Arms: Conservative Treatment

SUMMARY:
The purpose of this study is to create and test a treatment algorithm to guide the treatment of distal radius fractures in patients 65 and older and to obtain level-one evidence to determine the best method of treating distal radius fractures in this growing population demographic.

DETAILED DESCRIPTION:
* Distal radius fractures with borderline alignment will be randomized to surgical intervention or conservative treatment.
* Patients will fill out subjective questionnaires at 0, 6weeks, 3months, 6 months, and 1 year.
* Patients will perform objective strength tests, dexterity tests and have their range of motion tested at 12 weeks, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Distal Radius Fracture
* Between 10 and 20 degrees of dorsal angulation
* Between 3 and 5mm of Ulnar positive variance
* Between 1 and 2mm intra Articular Step deformity
* Age 65 and older

Exclusion Criteria:

* Pre-Morbid medical conditions which preclude surgical intervention
* Patients who do not live independently.
* Patients with an open fracture
* Associated soft tissue or skeletal injury to the same limb.
* Pre-existing wrist arthrosis or disability

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2008-11

PRIMARY OUTCOMES:
Primary: Patient pain and disability. Will be quantified with Disabilities of the Arm and Shoulder (DASH) and Patient Rated Wrist Evaluation (PRWE). | 0-1 year

SECONDARY OUTCOMES:
Secondary: To determine if other baseline factors influence outcome. For example, baseline activity levels (RAPA), home supports, hand dominance, and general mental health will be analyzed. | over 1 year
Secondary: To stratify results by age. (65-75, 77-80, and >80) | 0-1 year
Grip strength, Range of Motion and Dexterity testing of wrists | 3 months to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Joy C MacDermid, PhD, Principal Investigator — Hand and Upper Limb Centre, St. Joseph's Health Care; Ruby Grewal, MD, FRCSC, Principal Investigator — Hand and Upper Limb Centre, St Joseph's Health Care
Locations (2):
- Canada (2):
  - Hand and Upper Limb Centre, London, Ontario
  - Hand and upper Limb Centre, London, Ontario